CLINICAL TRIAL: NCT02318160
Title: Oxidative Status in Children and Adolescents With Autoimmune Thyroiditis: A Tertiary Center Study From Upper Egypt
Brief Title: Oxidative Status in Children With Autoimmune Thyroiditis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Saad, Associate professor of Pediatrics, Faculty of medicine,, Assiut University
Other Study IDs: AST123-2014
Record Dates: First submitted 2014-12-11; First posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Autoimmune Thyroiditis
Keywords: Autoimmune Thyroiditis; Oxidative Status; Children
MeSH Terms: conditions — Thyroiditis, Autoimmune

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: measurement of oxidant status in AIT — measurement of thyroid-stimulating hormone (TSH) and free thyroxin (FT4), as well as anti-thyroid peroxidase antibodies (TPOAb) and anti-thyroglobulin antibody (TgAb) were done in addition to assessment of malondialdehyde (MDA) and total antioxidant capacity (TAC) levels as an oxidative stress markers

SUMMARY:
Oxidative status in autoimmune thyroiditis was not investigated previously in children and adolescents. We investigated oxidant and antioxidant systems in a cohort of Egyptian children and adolescents with AIT to explore their relation with biomarkers of autoimmunity and thyroid function.

DETAILED DESCRIPTION:
Methods: A case control study included 32 children with autoimmune thyroiditis and 32 healthy subjects with matching age and sex were included as a control group. Thorough history, examination, thyroid ultrasound, measurement of thyroid-stimulating hormone (TSH) and free thyroxine (FT4), as well as anti-thyroid peroxidase antibodies (TPOAb) and anti-thyroglobulin antibody (TgAb) were done in addition to assessment of malondialdehyde (MDA) and total antioxidant capacity (TAC) levels as an oxidative stress markers. Results: Overt hypothyroidism was detected in 23/32 while subclinical hypothyroidism was detected in 9/32 of the studied patients. Malondialdehyde levels were significantly elevated while total antioxidant capacity levels were significantly decreased in autoimmune thyroiditis patients compared with healthy controls. The difference was more evident in patients with overt hypothyroidism than those with subclinical hypothyroidism. We also observed a significant positive correlation between anti-thyroid peroxidase antibodies levels and age, TSH, malondialdehyde, thyroid volume and a negative correlation with total antioxidant capacity and thyroxine .

Conclusions: The high serum malondialdehyde and lower total antioxidant capacity levels in patients with autoimmune thyroiditis and the correlation of thyroid antibodies with biomarkers of oxidative stress may reflect the role of autoimmunity in the development of oxidative stress. Future studies are needed for evaluation of the antioxidant therapy for autoimmune thyroiditis patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AIT.
* Age >6 years <18 years.
* Iodine sufficient region.

Exclusion Criteria:

* Children on antioxidants or antithyroid drugs
* Cardiac, renal and hepatic disease.
* Children with other autoimmune and collagen diseases

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Our case control study was conducted on 32 children and adolescents with Autoimmune Thyroiditis attending the Pediatric Endocrinology Clinic of Assiut University Children Hospital, Assiut, Egypt. . Diagnosis of Autoimmune Thyroiditis had been made by elevated anti-thyroid peroxidase antibodies (TPO Ab) and/or anti-thyroglobulin antibodies (Tg Ab) as well as typical hypoechogenicity of the thyroid in high-resolution sonography . Another group of 32 age and sex-matched healthy subjects as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Oxidative status | 3 months
  measurement of thyroid-stimulating hormone (TSH) and free thyroxine (FT4), as well as anti-thyroid peroxidase antibodies (TPOAb) and anti-thyroglobulin antibody (TgAb) were done in addition to assessment of malondialdehyde (MDA) and total antioxidant capacity (TAC) levels as an oxidative stress markers

REFERENCES:
- [Derived] Metwalley KA, Farghaly HS, Saad K, Othman HA. Oxidative status in children and adolescents with autoimmune thyroiditis. Clin Exp Med. 2016 Nov;16(4):571-575. doi: 10.1007/s10238-015-0386-x. Epub 2015 Sep 5. PMID 26343039